CLINICAL TRIAL: NCT02292823
Title: e-MASTER Registry: MGuard™ Prime Embolic Protection Stent in Patients With Acute ST Elevation Myocardial Infarction
Brief Title: MGuard™ Prime Embolic Protection Stent in Patients With Acute ST Elevation Myocardial Infarction
Acronym: e-MASTER
Status: Terminated | Type: Observational
Why Stopped: Enrolment rate
Sponsor: InspireMD (Industry)
Responsible Party: Sponsor
Other Study IDs: IMD-13
Record Dates: First submitted 2014-11-13; First posted 2014-11-17 (Estimated); Last update posted 2015-09-02 (Estimated); Status verified 2015-08

CONDITIONS: ST Elevation Myocardial Infarction
Keywords: STEMI; heart attack; stent; Bare Metal Stent; myocardial infarction; PCI
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Myocardial Infarction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: MGuard™ Prime Embolic Protection Stent System
  Other Names: MGuard™ Prime EPS

SUMMARY:
Prospective, non-randomized, single arm, multicenter observational study. The objective is to evaluate the safety and efficacy of the MGuard™ Prime stent in the treatment of de novo stenotic lesions in coronary arteries in patients undergoing primary percutaneous coronary intervention (PCI) due to acute ST elevation myocardial infarction (STEMI) in a real-world setting.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is >18 years of age.
2. Subject is experiencing clinical symptoms consistent with ST elevation acute myocardial infarction (STEMI) of >30 minutes and <24 hours.
3. Based on coronary anatomy, primary PCI is indicated for the culprit lesion with anticipated use of stenting.
4. Subject agrees to all required follow-up procedures and visits and has provided informed consent where required.
5. The target lesion is a de novo lesion in a native coronary artery.
6. The reference vessel diameter (RVD) of the infarct lesion is 2.75-4.0 mm by visual assessment.

Exclusion Criteria:

1. Subject undergoing cardiopulmonary resuscitation.
2. Cardiogenic shock (SBP <80 mmHg for >30 minutes, or requiring IV pressors or intra-aortic balloon bump (IABP) or other hemodynamic support device for hypotension).
3. Co-morbid condition(s) or others that could limit the subject's ability to participate in the trial or to comply with follow-up requirements, or impact the scientific integrity of the trial.
4. Target lesion involves a bifurcation with a side branch >/=2.0 mm in diameter.
5. In the Investigator's opinion the lesion/vessel is unsuitable for treatment with the MGuard™ Prime Embolic Protection Stent System for any reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects undergoing primary revascularization for STEMI and who are intended to undergo primary PCI with the MGuard™ Prime Embolic Protection Stent System.
Sampling Method: Non-Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2014-04; Primary Completion 2015-09 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Complete ST-segment resolution | 1 day
All cause death or MI at 30 days | 30 days

SECONDARY OUTCOMES:
TIMI flow grade | 1 day
Major Adverse Cardiac Events rate (MACE): cardiac death, re-MI, clinically-driven target lesion revascularization (TLR) | Discharge, 30 days, 6 months, 12 months
Acute success rates | 1 day
Stent thrombosis rate | Discharge, 30 days, 6 months,12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Onze Lieve Vrouwe Gasthuis, Amsterdam, Netherlands